CLINICAL TRIAL: NCT06779981
Title: A Prospective Epidemiological Cohort Study Evaluating Occurrences of Influenza-like Illness in an Urban Population of Healthy Subjects Aged 20-64 Years, Not Vaccinated Against Influenza.
Brief Title: A Prospective Epidemiological Study Evaluating Occurrences of Influenza-like Illness
Status: Completed | Type: Observational
Sponsor: Osivax (Industry)
Collaborators: Harmony Clinical Research BVBA (Other); Inferential (Industry); University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: OVX-FLU-002
Record Dates: First submitted 2025-01-14; First posted 2025-01-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Subjects experiencing influenza-like illness (ILI) symptoms will be asked to contact the investigational center to set up an additional visit within a maximum of 7 days of symptoms onset. During the additional visit, a nasopharyngeal swab will be collected to perform a reverse transcriptase-polymerase chain reaction (RT-PCR) assay to detect influenza A, influenza B, RSV, and/or SARS-CoV-2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective epidemiological cohort: Urban population of healthy subjects aged 20-64 years, not vaccinated against influenza.
  Interventions: Other: Nasopharyngeal swabs

INTERVENTIONS:
Other: Nasopharyngeal swabs — Completion of an electronic Diary (eDiary) and collection of nasopharyngeal swabs in case the subject experiences ILI symptoms
  Other Names: eDiary

SUMMARY:
This prospective epidemiological cohort study is being conducted in order to generate epidemiological data in support of Osivax's clinical development of a broad-spectrum influenza vaccine based upon the internal influenza nucleoprotein (NP), i.e., OVX836.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male or female participants, as determined by medical history and medical examination (as needed).
3. Between the ages of 20 and 64 years, inclusive.
4. Reliable and willing to make themselves available for the duration of the study, and willing and able to follow study procedures.
5. Ability and technical possibility for completing an eDiary.

Exclusion Criteria:

1. Subjects with a body mass index (BMI) ≤18 kg/m² or ≥35 kg/m²
2. Previous influenza vaccination within 6 months before the day of enrollment or planned to receive during the study duration.
3. Previous vaccination with an mRNA-based influenza vaccine including NP in its composition.
4. Previous administration of OVX836.
5. Pregnant or lactating woman.
6. Females planning to become pregnant or planning to discontinue contraceptive precautions until the end of the trial. Women of childbearing potential (WOCBP) should have appropriate contraceptive methods in place for 2 months before enrolment. Appropriate contraceptive methods are to be maintained until the end of the trial. Please also refer to Appendix A.
7. Past or current history of significant autoimmune diseases, as judged by the Investigator.
8. Current history of uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases.
9. Known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
10. Planned administration of any investigational or non-registered product during the entire study period.
11. History of receiving blood, blood components, or immunoglobulins within 3 months prior to the first study visit or planned to receive such product during the whole study period.
12. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
13. History of alcohol or drug abuse that ceased less than 6 months before enrolment, current alcohol or drug abuse according to the Investigator's judgement), smoking habit of more than 10 cigarettes/day, or current vaping (nicotine consumption corresponding to more than 10 cigarettes/day).
14. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months before the study vaccine administration. For corticosteroids, this will mean prednisone equivalent ≥20 mg/day. Inhaled, topical and intra-articular steroids are allowed.
15. Individuals with a history of any illness that, in the opinion of the Investigator, could potentially interfere with the results of the study or pose additional risk to the subjects by participating in the study.
16. Sponsor employees or Investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted, including children of newly composed families.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects, men and women aged 20 to 64 years.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants reporting ILI episodes (overall, laboratory confirmed or not), during the influenza season and during the whole study. | Through study completion, an average of 6 months.
Number and percentage of participants presenting RT-PCR confirmed influenza A or B cases, during the influenza season and during the whole study. | Through study completion, an average of 6 months.
Number and percentage of participants presenting RT-PCR confirmed SARS-CoV-2 cases, during the influenza season and during the whole study. | Through study completion, an average of 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Vaccinology (CEVAC), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No